CLINICAL TRIAL: NCT00349765
Title: Cardiovascular Health Effects of Isocaloric Substitution of Polyunsaturated Fat Rich Snacks for Saturated and Trans Fat or Refined Carbohydrate Snacks in Moderately Hypercholesterolemic Individuals.
Brief Title: Effects of Various Higher Fat and Lower Fat Snacks on Cardiovascular Risk Factors in Men and Women.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: SmartFoods, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: X041217008
Record Dates: First submitted 2006-06-30; First posted 2006-07-10 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Hypercholesterolemia
Keywords: cardiovascular disease; saturated fat; trans fat; polyunsaturated fat; diet; intramyocellular lipid
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: higher fat, high polyunsaturated fat diet
Behavioral: higher fat, high saturated and trans fat diet
Behavioral: lower fat diet

SUMMARY:
The purpose of this study is to determine whether snacks differing in fat amount and type result in changes in cardiovascular disease risk factors in men and women who have mildly elevated cholesterol levels. Our hypothesis is that a diet containing snacks rich in polyunsaturated fats lead to a more favorable cardiovascular disease risk profile than a diet containing snacks rich in saturated and trans fats or one containing low-fat snacks.

DETAILED DESCRIPTION:
The overall goals of this study are to determine whether snack foods rich in polyunsaturated fats (PUFA) produce beneficial effects on cardiovascular disease risk compared to snacks rich in saturated fats (SFA) and trans fats and snacks rich in refined carbohydrates. The primary objective of this study is to determine the effects of substituting n-6 PUFA (linoleic acid) from snack chips for SFA/trans fat and refined carbohydrate on serum lipids -principally LDL-C - and lipoproteins in moderately hypercholesterolemic men and women. A secondary objective is to assess effects on lipoprotein subclass particle size, intramyocellular lipids, and C-reactive protein (CRP). Forty-two men and women will be recruited to participate in a randomized, crossover, controlled feeding experiment for 3 periods of 4 weeks each. Each feeding phase will be separated by an 8-week washout period. The control diet will be a National Cholesterol Education Program Step 1 diet consisting of approximately 30% energy from total fat, <10% energy from SFA, 5% energy from PUFA, 15% energy from monounsaturated fatty acids (MUFA), 1% energy from trans fat, 55% energy from carbohydrates, and 15% energy from protein. To achieve an isocaloric substitution with PUFA, 300 kcal coming from low-fat, high-carbohydrate snacks will be removed from the Step 1 diet (NCEP diet) and replaced with 300 kcal of PUFA-rich snacks (LO diet). Similarly, 300 kcal from snacks rich in SFA/trans fat will replace the same 300 kcal from the high-carbohydrate from the Step 1 diet for the high SFA diet (SF diet). Subjects will consumed all foods provided by the GCRC and nothing else during each feeding phase. Breakfast and lunch meals will be consumed at the GCRC on weekdays and breakfast on Saturdays. All other meals will be packed and consumed at home. The primary study variable will be serum/plasma LDL-cholesterol. Secondary variables will include lipids and lipoproteins including total cholesterol (TC), HDL-cholesterol, VLDL-cholesterol, and triglycerides, and intramyocellular lipids. Exploratory variables will include assessment of lipid subclass particle size and CRP, a marker of systemic inflammation. Supportive variables will include fasting blood glucose and insulin, percent body fat mass, blood pressure and demographic information. All variables will be measured at baseline and endpoint of each feeding phase.

ELIGIBILITY:
Inclusion Criteria:

* age 19-65
* body mass index 20-35
* weight stable for at least 3 months
* low-density lipoprotein cholesterol 130-180 mg/dL
* triglycerides < 150 mg/dL
* glucose < 126 mg/dL

Exclusion Criteria:

* smokers
* type 1 diabetes
* type 2 diabetes
* use of lipid-lowering medications
* hypertension
* pregnancy
* lactation
* planning to become pregnant during the period of the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2005-03; Study Completion 2006-02

PRIMARY OUTCOMES:
total cholesterol
low-density lipoprotein cholesterol
high-density lipoprotein cholesterol
triglycerides

SECONDARY OUTCOMES:
C-reactive protein
lipoprotein a
very low-density lipoprotein cholesterol
LDL pattern A or B
blood pressure
body fat
waist circumference
intramyocellular lipid

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Result] St-Onge MP, Aban I, Bosarge A, Gower B, Hecker KD, Allison DB. Snack chips fried in corn oil alleviate cardiovascular disease risk factors when substituted for low-fat or high-fat snacks. Am J Clin Nutr. 2007 Jun;85(6):1503-10. doi: 10.1093/ajcn/85.6.1503. PMID 17556685